CLINICAL TRIAL: NCT01886690
Title: A Study to Compare the Safety and Efficacy of a New Eye Drop Formulation With REFRESH PLUS® in Participants Following LASIK Refractive Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11002X-002
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Bilateral LASIK Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Eye Drop Formulation (Experimental): 1 to 2 drops of carboxymethylcellulose sodium based New Eye Drop Formulation in each eye as per protocol for 90 days.
  Interventions: Drug: carboxymethylcellulose sodium based new eye drop formulation
- REFRESH PLUS® (Active Comparator): 1 to 2 drops carboxymethylcellulose sodium based (REFRESH PLUS®) eye drops in each eye as per protocol for 90 days.
  Interventions: Drug: carboxymethylcellulose sodium based eye drops

INTERVENTIONS:
Drug: carboxymethylcellulose sodium based new eye drop formulation — 1 to 2 drops of carboxymethylcellulose sodium based New Eye Drop Formulation in each eye as per protocol for 90 days.
  Arms: New Eye Drop Formulation
Drug: carboxymethylcellulose sodium based eye drops — 1 to 2 drops carboxymethylcellulose sodium based (REFRESH PLUS®) eye drops in each eye as per protocol for 90 days.
  Other Names: REFRESH PLUS®
  Arms: REFRESH PLUS®

SUMMARY:
This study will compare the safety and efficacy of a new eye drop formulation with REFRESH PLUS® in participants following LASIK surgery.

ELIGIBILITY:
Inclusion Criteria:

-Patients scheduled for LASIK surgery in both eyes.

Exclusion Criteria:

* Any systemic medication use within 3 months of screening (including over the counter, herbal, prescription, or nutritional supplement) which may affect dry eye or vision
* Use of topical eye medication other than prescribed for use in pre- or post-operative care
* Use of RESTASIS® or other topical ophthalmic cyclosporine product within 6 months prior to Screening
* Eye infection, inflammation, or allergy
* Soft contact lenses in the previous 7 days or rigid contact lenses in the previous 30 days prior to LASIK surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2014-08-18 (Actual); Study Completion 2014-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- New South Wales, Australia
- Kelowna, British Columbia, Canada

REFERENCES:
- [Background] Wallerstein A, Jackson WB, Chambers J, Moezzi AM, Lin H, Simmons PA. Management of post-LASIK dry eye: a multicenter randomized comparison of a new multi-ingredient artificial tear to carboxymethylcellulose. Clin Ophthalmol. 2018 May 7;12:839-848. doi: 10.2147/OPTH.S163744. eCollection 2018. PMID 29765198

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Eye Drop Formulation | REFRESH PLUS®
Started | 75 | 73
Completed | 75 | 71
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Personal Reasons | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Eye Drop Formulation | REFRESH PLUS® | Total
Number analyzed (Participants) | 75 | 73 | 148
Age, Customized [Number; unit: Participants]
  < 40 years | 58 | 51 | 109
  ≥ 40 years | 17 | 22 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 75
  Male | 39 | 34 | 73

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Disease Index© (OSDI) Score Using a 5-Point Scale
Description: The OSDI© is a 12-question survey for patients to document their dry eye disease symptoms. Each question is rated on a 5-point scale (0=none of the time and 4 = all of the time). The scores are totaled over the 12 questions and normalized/converted to a score of 0-100 (0=no disability and 100=complete disability).
Time Frame: Day 90
Population: Per Protocol: all randomized patients who had no significant protocol violations
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | New Eye Drop Formulation | REFRESH PLUS®
Number analyzed (Participants) | 68 | 57
Scores on a Scale | 6.99 (8.511) | 6.63 (7.071)

2. Secondary Outcome: Change From Baseline in Corneal Staining in the Worse Eye
Description: The cornea is the transparent front part of the eye which covers the iris and pupil. Corneal staining in the worse eye following administration of fluorescein dye in the eye is graded using a 6-point scale (0=no staining, 5=severe staining) over 5 areas of the clear central part of the eye for a minimum score of 0 and maximum score of 25. The higher the grade score, the worse the dry eye condition. A negative change from baseline represents a decrease in corneal staining (improvement) and a positive change from baseline represents an increase in corneal staining (worsening).
Time Frame: Baseline, Day 90
Population: Per Protocol: all randomized patients who had no significant protocol violations and who had data at the noted time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | New Eye Drop Formulation | REFRESH PLUS®
Number analyzed (Participants) | 68 | 58
Scores on a Scale
  Baseline | 0.9 (1.28) | 1.2 (1.31)
  Change from Baseline at Day 90 (N=68, 57) | 0.2 (1.96) | -0.3 (1.61)

3. Secondary Outcome: Change From Baseline in Tear Break-up Time (TBUT) in the Worse Eye
Description: TBUT is the time required for dry spots to appear on the surface of the eye after blinking in the worse eye. The longer it takes, the more stable the tear film. A short TBUT is a sign of poor tear film. A positive number change from baseline indicates an increase in TBUT (improvement) and a negative number change from baseline indicates a decrease in TBUT (worsening).
Time Frame: Baseline, Day 90
Population: Intent-to-Treat: all randomized patients who had data at the noted time point
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | New Eye Drop Formulation | REFRESH PLUS®
Number analyzed (Participants) | 75 | 73
Seconds
  Baseline | 11.88 (11.656) | 9.27 (5.121)
  Change from Baseline at Day 90 (N=75, 71) | 1.21 (9.299) | 1.08 (5.304)

4. Secondary Outcome: Change From Baseline in the Schirmer Test in the Worse Eye
Description: The Schirmer's Test measures the rate of the secretion of tears produced by the eye over 5 minutes in the worse eye. The results indicate the presence of dry eye (Normal = greater than or equal to 10 millimeters (mm) of tears, Dry Eye = less than 10 mm of tears). The smaller the number, the more severe the dry eye. A positive number change from baseline indicates an increase in tears (improvement) and a negative number change from baseline indicates a decrease in tears (worsening).
Time Frame: Baseline, Day 90
Population: Intent-to-Treat: all randomized patients who had data at the noted time point
Measure: Mean (Standard Deviation); unit: Millimeters in 5 minutes (mm/5 min)
Arm/Group | New Eye Drop Formulation | REFRESH PLUS®
Number analyzed (Participants) | 75 | 73
Millimeters in 5 minutes (mm/5 min)
  Baseline | 13.1 (9.10) | 13.0 (8.74)
  Change from Baseline at Day 90 (N=75, 71) | 1.4 (8.55) | 1.3 (9.89)

5. Secondary Outcome: Change From Baseline in Uncorrected Visual Acuity in the Worse Eye
Description: Uncorrected visual acuity in the worse eye is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) without corrective lenses. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive number change from baseline in the number of letters read correctly indicates an improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Letters Read Correctly
Arm/Group | New Eye Drop Formulation | REFRESH PLUS®
Number analyzed (Participants) | 68 | 58
Letters Read Correctly
  Baseline | 51.1 (10.00) | 53.1 (9.49)
  Change from Baseline at Day 90 (N=68, 57) | 5.8 (5.24) | 4.7 (6.02)

ADVERSE EVENTS:
Description: The Safety Population included all treated patients and was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | New Eye Drop Formulation | REFRESH PLUS®
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/73
Other Adverse Events (participants affected / at risk) | 4/75 | 18/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Eye Drop Formulation (N=75) | REFRESH PLUS® (N=73)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New Eye Drop Formulation (N=75) | REFRESH PLUS® (N=73)
Nasopharyngitis (Infections and infestations) | 2 | 4
Headache (Nervous system disorders) | 1 | 8
Blepharitis (Eye disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.